CLINICAL TRIAL: NCT05597761
Title: Immunogenicity of COVID-19 Vaccination in Immunocompromised Patients (Auto-COVID-VACC)
Status: Active, not recruiting | Type: Observational
Sponsor: Oliver Cornely, MD (Other)
Collaborators: ZKS Köln (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Oliver Cornely, MD, Principal Investigator, University of Cologne
Organization: University of Cologne (Other)
Other Study IDs: AUTO-COVID-VACC-4943
Record Dates: First submitted 2022-10-26; First posted 2022-10-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-11

CONDITIONS: COVID-19; Adult; Immunocompromised Patients
Keywords: COVID-19; mRNA vaccination; Immunocompromised patients
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This multicenter, prospective, non-interventional study aims to evaluate data on humoral and cellular immune response generated within the COVID-19 vaccination standard in immunocompromised patients.

DETAILED DESCRIPTION:
This study aims to analyze the immune response data generated within the procedures of the standard-of-care COVID-19 vaccination. for immunocompromised patients.

Additional blood will be drawn from the patients at each visit defined within the vaccination standard by using the same vein puncture as used for blood drawings of routine blood samples. Study related blood samples will be used for evaluation of T and B cell response to COVID-19 vaccinations.

For this study, no additional visits or invasive procedures will be performed in addition to the standard interventions.

ELIGIBILITY:
Inclusion criteria:

* Patient is vaccinated according to the recent version of the COVID-19 vaccination standard for immunocompromised patients.
* Patient is 18 years of age or older at enrollment.
* Written informed consent from patient has been obtained prior to any study related procedures

Exclusion criteria:

• Patient is not vaccinated according to the recent version of the COVID-19 vaccination standard. Patient has a positive SARS-CoV-2 antigen test at the first visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Immunocompromised patients
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anti-Spike-IgG titers | At the end of each vaccination cycle (each cycle is 28 days)
  Time to an adequate immune response according to the recent version of the COVID-19 vaccination standard after repeated mRNA vaccinations

SECONDARY OUTCOMES:
BA.1-specific neutralizing antibody ID50 titers | At the end of each vaccination cycle (each cycle is 28 days)
  Time to Omicron BA.1-specific neutralizing antibody ID50 titers ≥20/ml after repeated mRNA vaccinations
Anti-Spike-1/2 IgG increase >33.8 BAU/ml | At the end of each vaccination cycle (each cycle is 28 days)
  Time to anti-Spike-1/2 IgG increase >33.8 BAU/ml after repeated mRNA vaccinations in immunocompromised patients
Decrease of BA.1-specific neutralizing antibody ID50 titers | Every 28 days following last COVID-19 vaccination for a total duration of 24 weeks
  Time to decrease of Omicron BA.1-specific neutralizing antibody ID50 titers <20/ml after last mRNA vaccine in successfully vaccinated patients
Anti-Spike-1/2 IgG decrease ≤33.8 BAU/ml | Every 28 days following last COVID-19 vaccination for a total duration of 24 weeks
  Time to anti-Spike-1/2 IgG decrease ≤33.8 BAU/ml after last mRNA vaccine in successfully vaccinated patients

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A. Cornely, Prof., Principal Investigator — University Hospital of Cologne, Internal Medicine I
Locations (3):
- Germany (3):
  - Klinik für Hämatologie, Onkologie, Hämostaseologie und Stammzelltransplantation (Med. Klinik IV) Uniklinik der RWTH Aachen, Aachen, North Rhine-Westphalia
  - University Hospital of Cologne, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Essen Klinik für Hämatologie und Stammzellentransplantation, Essen, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cremer LM, Bethe U, Borchmann P, Di Cristanziano V, Gieselmann L, Grimm S, Hellmich M, Jakobs J, Nacov JA, Neuhann JM, Prattes J, Scheid C, Sprute R, Steger G, Stemler J, Mellinghoff SC, Cornely OA. Immunogenicity of COVID-19 Vaccination in Immunocompromised Patients (Auto-COVID-VACC): Protocol for Multicenter Prospective Noninterventional Study. JMIR Res Protoc. 2025 May 26;14:e60675. doi: 10.2196/60675. PMID 40418566